CLINICAL TRIAL: NCT06468124
Title: Prospective Study to Correlate the Treatment Sensitivity of Patient-derived Organoids With Clinical Outcomes in Breast Cancer Patients With Brain and/or Extra-cranial Metastases
Brief Title: Sensitivity of Organoids to Predict Treatment Outcome in Breast Cancer Metastases
Acronym: PDO
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 315793
Record Dates: First submitted 2024-06-04; First posted 2024-06-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Tumour and normal tissues, blood, saliva, oral swabs, urine and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer patients with brain metastases: Breast cancer patients with brain metastases undergoing surgical resection with or without further radiotherapy (SRS or whole brain radiotherapy)
- Breast cancer patients with extra-cranial metastases: Breast cancer patients with extra-cranial metastases undergoing surgical resection or biopsy

SUMMARY:
The aim of the study is to generate patient-derived organoids (PDOs) from brain resection or biopsied extra-cranial metastases. The preliminary data collected will be used to assess the ability of PDOs to predict patients' treatment response and their radio-sensitivity and chemo-sensitivity can be correlated with their survival outcome.

DETAILED DESCRIPTION:
The SOTO-BC trail is an observation study and the patients will continue their clinical visits and follow-up as per normal standard of care.

Patient cohorts:

1. Breast cancer patients with brain metastases undergoing surgical resection with or without further radiotherapy (SRS or whole brain radiotherapy)
2. Breast cancer patients with extra-cranial metastases undergoing surgical resection or biopsy

Primary objective:

To assess the percentage of successful generated organoids from resected brain or resected/biopsied extra-cranial metastases of breast cancer patients

Secondary objectives:

1. To assess the sensitivity of radiotherapy in PDOs
2. To assess the sensitivity of the same systemic treatments that the patients previously had and will have in PDOs
3. To correlate the treatment sensitivities of PDOs above with the treatment outcome of patients
4. To correlate IC50 doses/dose response curves above with the objective response rates of patients undergoing same systemic treatment

Study Procedures:

Breast cancer patients with resectable brain or extra-cranial metastases or who will undergo a biopsy of the extra-cranial metastases will be asked to consent for this study and for their resected/biopsied samples to be used to generate PDOs. The investigators aim to recruit 20 patients in the pilot phase of the study.

When the PDOs contain sufficient cells, these cells will be treated with increasing doses of radiotherapy and/or relevant systemic treatments in order to determine the IC50 and to obtain dose-response curves of these PDOs to the treatments. The investigators will treat the PDOs with the same treatments that the patients had or will receive in order to correlate the responses to radiotherapy and/or systemic treatments including immunotherapy (co-cultured with immune cells).

The response of these PDOs will be compared to the treatment outcome and survivals in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with brain metastases who are suitable for surgical resection or Breast cancer patients with extra-cranial metastases undergoing surgical resection or biopsy
* Age > 18 years old

Exclusion Criteria:

* Patients unable to give informed consent e.g., mental disability or vulnerable adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with resectable brain or extra-cranial metastases and undergoing postoperative radiotherapy or palliative radiotherapy to extracranial metastases if necessary +/- other systemic treatments after resection. Patients who will undergo a biopsy of the extra-cranial metastases may be recruited and asked to consent for an additional research biopsy at the same time as standard of care biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient derived organoids | 10 months
  To generate PDOs from brain or extra-cranial metastases of breast cancer patients.

SECONDARY OUTCOMES:
Response to radiotherapy | 6 months
  To determine the dose response curves of radiotherapy
Response to therapy | 5 months
  To determine the IC50 doses of the previous and same systemic treatments that patients had or will have in PDOs
recurrence and survival rates | 4 months
  To correlate the IC50 doses and dose response curves above with the recurrence rates and progression-free survival of patients
Response rate of patients undergoing systemic treatment | 3 months
  To correlate IC50 doses/dose response curves above with the objective response rates of patients undergoing same systemic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kong, Principal Investigator — Clinical reader and honorary NHS consultant in clinical oncology
Locations (2):
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT06468124/Prot_000.pdf